CLINICAL TRIAL: NCT03415165
Title: Efficacy of 200mg and 300mg Concentrates of Green Tea Polyphenols Using Buccal Tablets Versus Topical Application of Corticosteroids in Treatment of Patients With Symptomic Oral Lichen Planus Randomized Clinical Trial
Brief Title: Efficacy of Green Tea Buccal Tablets in Oral Lichen Planus
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Magdy, princible investigator EMagdy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 161187
Record Dates: First submitted 2018-01-22; First posted 2018-01-30 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- green tea buccal tablet (Active Comparator): buccal tablet 3 times aday
  Interventions: Drug: green tea buccal tablet
- corticosteroids topical (Sham Comparator): topical steroids 3 times aday
  Interventions: Drug: Corticosteroids Topical

INTERVENTIONS:
Drug: green tea buccal tablet — buccal tablet for 8 hrs 3 times aday
  Other Names: catechines
  Arms: green tea buccal tablet
Drug: Corticosteroids Topical — kenacort in orabase 4 times aday
  Other Names: local corticosteroids
  Arms: corticosteroids topical

SUMMARY:
Is topical application of green tea polyphenols buccal tablet more effective in treatment of patients with symptomatic oral lichen planus in comparison with topical application of corticosteroids and what is the most effective concentration of polyphenols

DETAILED DESCRIPTION:
* Each patient was informed about the detailed procedure, and educated about benefits of the treatment, the known side effects and follow-up appointments needed. After that, each subject participating in the study signed an informed written consent form.
* Subjects were given freedom to leave the study at any time when they need to. Group A (Experimental group) 200 mg green tea

Where patients in this group will receive a buccal tablet containing 200 mg of green tea extract which adheres to the buccal mucosa slowly releasing the polyphenoles along around 8 hours 2 times aday for four weeks.

Preparation of buccal tablets : Mucoahesive buccal tablets is prepared by a direct compression procedure. Various batches are prepared by varying the chitosan:drug ratio to identify the most effective formulation. The mucoadhesive drug/polymer mixture is prepared by homogeneous mixing of the drug with chitosan , secondary polymer, and D-mannitol, in a glass mortar for 15 min. Then, Mg stearate will be added and mixed for 5 min .The mixture is compressed using a tablet machine (Type EK: O.Erweka apparatus, Frankfurt, Germany) using flat-tip punches and dies with 8-mm-diameter. Each tablet weighed 212 mg with a thickness of 3.1 mm.( Darwish and Elmeshad,2009)

Group B (Experimental group) 300 mg green tea

Where patients in this group will receive a buccal tablet containing 300 mg of green tea extract which adheres to the buccal mucosa slowly releasing the polyphenoles along around 8 hours 2 times aday for four weeks.

Group C (Control group) corticosteroid group:

Where patients are treated with topical corticosteroids 1 mg/g Triamcinolone acetonide (Kenacort-A orabase 20 G Pomad: Deva dermatological product,Turkey) applied topically 4 times a day i.e. following each meal and at bed time for four weeks .

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic lesions.
* OLP lesions with the diagnosis confirmed both clinically and histopathologically.
* Clinical score higher than 3.
* Disease duration of more than 2 months.
* Absence of dysplasia in histological section

Exclusion Criteria:

* Presence of any visible oral lesion other than OLP.
* Pregnant or breast-feeding women,
* Immuno-deficiency diseases.
* Current malignancy or malignancy in history.
* Concomitant treatment potentially effective on OLP within the previous 2 months such as antimalarial agents, retinoids, corticosteroids or immunosuppressive drugs.
* Severe or recurrent infections.
* Lichenoid reaction.
* Patients presents with skin lesions which may require systemic corticosteroid therapy.

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
size of the lesion | 12 weeks
  the shape and the measurement of its size

SECONDARY OUTCOMES:
visual analogue score | 12 weeks
  pain score from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: cairo university, Study Chair — cu
Locations (1):
- Cairo University, Cairo, Egypt